CLINICAL TRIAL: NCT05215015
Title: Clinical Study of Conjugated Antibody Redirecting Natural Killer (CAR-NK) Cells Targeting CD33 and CLL1 in Patients With Acute Myeloid Leukemia
Brief Title: Study of Anti-CD33/CLL1 CAR-NK in Acute Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Collaborators: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBR733-T01; WX-IBR-7 (Other: Wuxi People's Hospital)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD33/CLL1 CAR-NK Cells (Experimental): The administration of CAR-NK cells will be performed on day 1 and day 3 of each cycle (28 days). The first administration dose in the first cycle is 2.0×10^9 cells. If no adverse events were observed, the second administration dose in the first cycle would be 3.0×10^9 cells, and each administration dose in the second cycle and thereafter would be 3.0×10^9 cells.
  Interventions: Biological: Anti-CD33/CLL1 CAR-NK Cells

INTERVENTIONS:
Biological: Anti-CD33/CLL1 CAR-NK Cells — The administration of CAR-NK cells will be performed on day 1 and day 3 of each cycle (28 days). The first administration dose in the first cycle is 2.0×10^9 cells. If no adverse events were observed, the second administration dose in the first cycle would be 3.0×10^9 cells, and each administration dose in the second cycle and thereafter would be 3.0×10^9 cells.

SUMMARY:
This is an open-label, nonrandomized, investigator-initiated clinical trial to evaluate the safety, tolerability, pharmacokinetics, and efficacy of anti-CD33/CLL1 CAR-NK cell injection in patients with acute myeloid leukemia (AML), and to determine PK parameters, maximum tolerated dose (MTD), and phase II recommended dose (RP2D) for subjects receiving CAR-NK cell injection.

DETAILED DESCRIPTION:
The treatment cycle in this study is 28 days. The administration of CAR-NK cells will be performed on day 1 and day 3 of each cycle. Subjects will be treated continuously until the criteria for termination of treatment are met. In this study, the dose escalation design is adopted. The first administration dose in the first cycle is 2.0×10^9 cells. If no adverse events were observed, the second administration dose in the first cycle would be 3.0×10^9 cells, and each administration dose in the second cycle and thereafter would be 3.0×10^9 cells.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should voluntarily participate in this clinical study, are fully aware of the study, have signed the Informed Consent Forms, and are willing to follow and able to complete all trial procedures.
2. Subjects who are more than 18 years old (including 18 years old), and less than 75 years old (including 75 years old);
3. Subjects who are diagnosed as AML according to the World Health Organization (WHO) 2016 diagnosis criteria, and meet any of the following:

   * Relapsed acute myeloid leukemia: after complete response (CR), there are leukemia cells in peripheral blood or blast cells in bone marrow >5% (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration.
   * Refractory acute myeloid leukemia: treatment-naive subjects who have no response to the standard of care for 2 courses of treatment; subjects who are relapsed within 12 months with consolidated intensive treatment after CR; subjects who are relapsed after 12 months but have no response to the conventional chemotherapy; subjects who are relapsed twice or more; subjects who have persistent extramedullary leukemia.
4. Subjects who are positive in CD33 or CLL1 test (according to the results of the central laboratory);
5. Subjects are allowed to have received ≤1 autologous HSCT;
6. Subjects whose performance status scores of the Eastern Cooperative Oncology Organization (ECOG) are≤2;
7. Subjects with the expected survival phase>3 months;
8. Organ function should meet the following criteria:

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN), unless these are caused by leukemia cell infiltration as determined by the investigator;
   * Total serum bilirubin ≤ 1.5 times the upper limit of normal (ULN);
   * Glomerular filtration rate (GFR)>50 mL/min;
   * Left ventricular ejection fraction (LVEF)≥50%, no clinically significant pericardial effusion confirmed by echocardiography;
   * Blood oxygen saturation under indoor ventilation in the screening phase>92%;
9. Female subjects of childbearing age must be negative in the pregnancy test results in the screening phase;
10. Male and female subjects of childbearing age must agree to take effective birth controls after signing the informed consent forms, during the study, and within 6 months after the last administration.

Exclusion Criteria:

1. Subjects who are known to have acute promyelocytic leukemia;
2. Subjects who suffer from or are suspected of suffering from central nervous system leukemia, or central nervous system involvement;
3. Subjects who have received allogeneic HSCT;
4. Subjects who have prior II-IV (Glucksberg criteria) acute graft versus-host disease (GvHD) or extensive chronic GvHD;
5. Subjects who have received chimeric antigen receptor cell therapy or other cell therapy;
6. Subjects who have received anti-tumor therapy in the early stage but are not recovered in the toxicity (according to NCI-CTCAE 5.0, the toxicity has not recovered to ≤ Grade 1, except for fatigue, anorexia, and alopecia);
7. Subjects who have had other malignant tumors within 5 years before inclusion, except for any type of carcinoma in situ that has been cured in the past and cured skin basal cell carcinoma or skin squamous cell carcinoma;
8. Subjects whose cardiac function and disease meet one of the following conditions within 6 months before the first administration:

   * Any risk factors that increase QTcF (Fridericia formula) interval prolongation, such as uncorrectable hypokalemia, hereditary long QT syndrome, and use of drugs that prolong the QTcF interval;
   * New York Heart Association (NYHA) classification ≥Grade 3;
   * QTcF interval prolongation (male>450 milliseconds; female>470 milliseconds);
   * Unstable angina pectoris, and myocardial infarction;
9. Subjects who have a history of autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.) that require systemic immunosuppressive/systemic disease modulating drugs within 2 years before the first administration;
10. Subjects who have active systemic fungal, bacterial or viral infections that are uncontrolled or are required to be treated by intravenous administration;
11. Subjects with human immunodeficiency virus (HIV) antibody positive;
12. Subjects with HBsAg (-) and HBcAb (-). If subjects have HBsAg (+) and/or HBcAb (+), then subjects with HBV-DNA below the local lower limit of quantification can be included;
13. Subjects with hepatitis C virus antibody (-). If subjects have hepatitis C virus antibody (+), then subjects with HCV-RNA (-) can be included;
14. Female subjects who are breastfeeding and unwilling to stop breastfeeding;
15. Subjects who have received major surgery (for the definition of major surgery, refer to the Level 3 and 4 surgeries specified in the Administrative Measures for the Clinical Application of Medical Technology) within 28 days before the first administration.
16. Subjects who have received a solid organ transplant;
17. Subjects who have a history of alcohol, drug use or drug abuse;
18. Subjects who are known to be allergic to the study drug and/or main components and/or any excipients of the study drug;
19. Subjects who have other severe, acute, or chronic diseases or laboratory abnormalities that may increase the risk of participating in the study and receiving the study drug, or may interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | 28 days after initial infusion
  To evaluate the safety and tolerability of Anti-CD33/CLL1 CAR-NK cells

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 1 year after infusion
  To evaluate the effectivity of anti-CD33/CLL1 CAR-NK cells
Minimal residual disease (MRD) | Up to 1 year after infusion
  To evaluate the effectivity of anti-CD33/CLL1 CAR-NK cells
Objective response rate (ORR) | Up to 1 year after infusion
  To evaluate the effectivity of anti-CD33/CLL1 CAR-NK cells
Duration of overall response (DOR) | Up to 1 year after infusion
  To evaluate the effectivity of anti-CD33/CLL1 CAR-NK cells
Plasma concentration of CAR-NK cells | One month after the last infusion
  Blood samples will be collected at specified time points to detect the number of CAR-NK cells in peripheral blood and to evaluate the PK parameters
Cytokine release | One month after the last infusion
  Blood samples will be collected at specified time points to detect the cytokine (IL-6, TNF-α, IL-1ra, IL-10, IL-2, etc.) concentration (pg/mL)
Adverse Events (AEs) | From day 1 to day 90 after the last infusion
  The incidence and severity of adverse events assessed according to Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, and the correlation between adverse events and CAR-NK cells
Percentage of subjects receiving hematopoietic stem cell transplantation (HSCT) | Up to 1 year after infusion
  To explore HSCT in subjects receiving CAR-NK cell therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No